CLINICAL TRIAL: NCT06988722
Title: Comparative Effects of 650 nm and 810 nm Diode Laser Photobiomodulation on Postoperative Pain, Analgesic Use, and OHRQoL After Dental Implant Surgery: A Randomized Controlled Trial
Brief Title: Laser Photobiomodulation After Dental Implant Surgery: A Comparison of 650 nm and 810 nm Diode Lasers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Laser Enhanced Sciences (Other)
Responsible Party: Principal Investigator, Dr. Mohammad Mahmoud Yehya Abdussalam, Principal Investigator, National Institute of Laser Enhanced Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZZA-PBM-2024-RCT01; NILES-EC-CU 23/7/18(In) (Other: NILES, Cairo University)
Record Dates: First submitted 2025-05-14; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Postoperative Pain; Dental Implant
Keywords: Photobiomodulation; Low-Level Laser Therapy; Diode Laser; 650 nm Laser; 810 nm Laser; Dental Implant Surgery; Pain Management; OHIP-14; OHRQoL; Numerical Rating Scale
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Participants were randomized into three groups: 650 nm PBM, 810 nm PBM, or sham laser therapy. Each group received only one type of intervention.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessors were blinded to group allocation. The operator administering the laser therapy was not blinded due to the nature of the device used. Sham PBM was visually identical to active laser settings to maintain blinding for all other parties.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 650 nm PBM (Experimental): Participants in this arm received photobiomodulation therapy using a 650 nm red diode laser. The laser was applied at three points (buccal, palatal, and crestal) around the implant site at 100 mW for 60 seconds per point, delivering a total dose of 18 J. PBM was applied immediately after implant placement and repeated within 48 hours.
  Interventions: Device: 650 nm Diode Laser PBM
- 810 nm PBM (Experimental): Participants in this arm received photobiomodulation therapy using an 810 nm infrared diode laser. The laser was applied at three points (buccal, palatal, and crestal) around the implant site at 100 mW for 60 seconds per point, delivering a total dose of 18 J. PBM was applied immediately after implant placement and repeated within 48 hours.
  Interventions: Device: 810 nm Diode Laser PBM
- Sham PBM (Sham Comparator): Participants in this arm received sham photobiomodulation therapy. The same laser handpiece was applied at the same points and durations as the active groups, but with the laser emission disabled. The procedure was designed to appear identical to active PBM treatment to maintain blinding. The sham was applied immediately after implant placement and repeated within 48 hours.
  Interventions: Device: Sham Laser PBM

INTERVENTIONS:
Device: 650 nm Diode Laser PBM — A 650 nm red diode laser applied at three points (buccal, palatal, and crestal) around the implant site using 100 mW power for 60 seconds per point (total dose 18 J). Applied immediately post-op and repeated within 48 hours. Used for photobiomodulation to reduce pain and improve healing.
  Other Names: Red laser therapy; Low-Level Laser Therapy (650 nm)
  Arms: 650 nm PBM
Device: 810 nm Diode Laser PBM — A 810 nm red diode laser applied at three points (buccal, palatal, and crestal) around the implant site using 100 mW power for 60 seconds per point (total dose 18 J). Applied immediately post-op and repeated within 48 hours. Used for photobiomodulation to reduce pain and improve healing.
  Other Names: Infrared laser therapy; Low-Level Laser Therapy (810 nm); Near-Infrared laser therapy
  Arms: 810 nm PBM
Device: Sham Laser PBM — Identical laser handpiece applied at the same locations and durations as the active PBM groups, but without laser emission. Used to maintain blinding and simulate treatment without therapeutic effect.
  Other Names: Sham Photobiomodulation; Inactive Laser
  Arms: Sham PBM

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of laser light therapy, known as photobiomodulation (PBM), in reducing pain after dental implant surgery. The study involves adult patients receiving a single dental implant in the upper posterior (back) area of the mouth. Participants are randomly assigned to receive PBM using either a 650 nm red diode laser, an 810 nm infrared diode laser, or a sham (inactive) laser.

The study aims to assess whether PBM therapy can reduce pain during the first three days after surgery, decrease the need for pain medication, and improve oral health-related quality of life (OHRQoL). PBM is applied immediately after surgery and again within 48 hours. Pain intensity is measured at multiple time points (2, 6, 12, 24, 48, and 72 hours), analgesic use is recorded, and OHRQoL is evaluated using a standardized questionnaire.

DETAILED DESCRIPTION:
This randomized, double-blind, sham-controlled clinical trial assessed the short-term effects of photobiomodulation (PBM) using 650 nm and 810 nm diode lasers on postoperative pain, analgesic intake, and oral health-related quality of life (OHRQoL) following single dental implant placement in the posterior maxilla.

Methods:

Sixty participants were randomized into three equal groups (650 nm PBM, 810 nm PBM, or sham). All underwent a standardized H-design flap surgery and implant placement. PBM was applied at three points around the implant (buccal, palatal, crestal) using 100 mW power for 60 seconds per point (total 18 J), repeated within 48 hours.

Outcomes:

Primary outcome: Pain intensity measured using an 11-point Numeric Rating Scale (NRS) at 2, 6, 12, 24, 48, and 72 hours after surgery.

Secondary outcomes: Number of analgesics used (acetaminophen 1000 mg as needed), and changes in OHRQoL as measured by the OHIP-14 questionnaire at baseline, 1 week after implant placement, and 1 week after crown delivery.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20-65 years.
* Indicated for single dental implant placement in the posterior maxilla.
* ASA physical status I or II.
* Good oral health.
* Willingness and ability to comply with study procedures and follow-up schedule.
* Able to provide written informed consent.

Exclusion Criteria:

* Use of analgesics, NSAIDs, or corticosteroids within 48 hours prior to surgery.
* History of alcohol abuse or regular consumption of >14 drinks/week (men) or >7 drinks/week (women), or withdrawal within the last 6 months.
* History of chronic pain or long-term pain medication use.
* Need for grafting, sinus lift, or complex implant procedures.
* Pregnant or breastfeeding.
* Uncontrolled systemic disease (e.g., uncontrolled diabetes, immunodeficiency).
* History of epilepsy, photosensitivity, or contraindications to laser therapy.
* Allergy or contraindication to acetaminophen.
* Previous implant or surgical treatment in the same site within the past 6 months.
* Heavy smokers (>12 cigarettes/day) or individuals who quit smoking within the past 6 months.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-08-17 (Actual); Primary Completion 2024-06-02 (Actual); Study Completion 2024-06-29 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Intensity Using Numeric Rating Scale (NRS) | 2, 6, 12, 24, 48, and 72 hours after surgery
  Postoperative pain intensity was assessed using an 11-point Numeric Rating Scale (NRS: 0-10) at 2, 6, 12, 24, 48, and 72 hours after surgery. Participants recorded the maximum pain experienced since the previous interval. Pain was analyzed in two ways: (1) Temporal analysis of mean NRS scores across Day 1 (defined as the highest score within 24 hours), Day 2, and Day 3 to assess daily pain evolution; and analysis of specific time points on Day 1 (2, 6, 12, 24 hours) to explore early postoperative pain dynamics. (2) Categorical analysis of NRS scores classified into five pain severity levels: no, mild, moderate, severe, and unbearable pain. Group comparisons were conducted using ANOVA or Kruskal-Wallis tests for continuous data and Chi-square tests for categorical distributions.

SECONDARY OUTCOMES:
Analgesic Intake (Acetaminophen 1000 mg) | 2, 6, 12, 24, 48, and 72 hours after surgery
  Analgesic use was self-recorded at 2, 6, 12, 24, 48, and 72 hours postoperatively. At each interval, participants documented whether they had taken a 1000 mg dose of acetaminophen within the prior 4 hours (Yes/No). This binary outcome was used to correlate pain scores with analgesic consumption and to assess the frequency of rescue medication use across study groups. Participants were instructed to take acetaminophen only if their pain exceeded an NRS score of 3.
Oral Health-Related Quality of Life (OHRQoL) Using OHIP-14 | Baseline, 1 week post-implant placement, and 1 week post-prosthesis placement
  OHRQoL was measured using the validated Oral Health Impact Profile-14 (OHIP-14) questionnaire. Participants completed the OHIP-14 electronically at three time points: baseline (before surgery), 1 week after implant placement, and 1 week after prosthesis placement. The impact of treatment on oral health-related quality of life was evaluated by comparing OHIP-14 scores within and between groups over time.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad M Abdussalam, BDS, MSc, Principal Investigator — National Institute of Laser Enhanced Sciences (NILES), Cairo University
Locations (1):
- National Institute of Laser Enhanced Sciences (NILES), Cairo University, Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in this article will be made available after de-identification, upon reasonable request and following institutional and ethical approvals. Supporting documents such as study protocol and statistical analysis plan may also be shared as needed.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be shared beginning 6 months following publication and will be available for up to 3 years upon reasonable request.
Access Criteria: * Data will be made available to qualified researchers for individual participant meta-analysis or academic research focused on dental implant outcomes and photobiomodulation. Requests should be submitted with a brief research proposal and data use agreement. Approved data will be shared electronically via email or a secure cloud-based system.
  * Mechanism of access: Requests should be sent to std.zein.adham@niles.edu.eg